CLINICAL TRIAL: NCT01352455
Title: A Pilot Study of More Frequent In-Center Hemodialysis to Improve Outcomes in Pediatric End Stage Renal Disease
Brief Title: More Frequent In-Center Hemodialysis in Pediatric End Stage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0596
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Pediatric End Stage Renal Disease; Hemodialysis
Keywords: Hemodialysis; Pediatric; Outcomes; Comparative Effectiveness; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5 days per week hemodialysis (Experimental): 5 days per week, 2 hours 20 minutes per session versus 3 days per week, 4 hours per session
  Interventions: Procedure: Hemodialysis

INTERVENTIONS:
Procedure: Hemodialysis — 5 days per week hemodialysis

SUMMARY:
A health kidney works 24 hours a day, 7 days a week to remove toxins and fluid from the body. Many children with permanent kidney failure undergo dialysis, a life saving procedure that takes the place of a kidney. Currently, many children with permanent kidney failure only receive dialysis treatments 3 days a week in the hospital dialysis clinic. Children on dialysis have a markedly reduced life expectancy, with a life span 40-50 years shorter than their healthy counterparts. Survival for these children has not improved over the last 20 years. These data indicate that the current dialysis treatment strategy is unacceptable.

This research project will study if more frequent dialysis, performed 5 days per week, will improve the health of children with permanent kidney failure compared to the current treatment strategy. Children will be treated with both traditional and more frequent dialysis schedules to measure improvements in their health and well being.

ELIGIBILITY:
Inclusion Criteria:

* Current outpatient ESRD pediatric patients, 3-21 years old, receiving in-center chronic HD.
* Patients have to be on chronic HD for at least 2 months before eligibility

Exclusion Criteria:

* Patients with a scheduled (with a specific transplant date) kidney transplant in the next 6 months
* Patients scheduled to be switched to peritoneal dialysis in the next 6 months
* Patients currently receiving >3 days per week of hemodialysis
* Patients currently receiving >12 hours per week of hemodialysis
* Anyone <3 years of age would be excluded from the study, so our minimum anticipated patient weight would be about 11 kg
* Patients >21 years of age at enrollment
* Patients receiving concomitant peritoneal dialysis
* Patients with <2 months on chronic HD
* Patients with a temporary or femoral dialysis catheter
* Patients who are not hypertensive (both not on blood pressure medication and with a SBP <95th percentile for age, sex, and height)
* Patients enrolled in an investigational drug trial involving blood pressure medication or any other clinical trial potentially affecting the primary outcome of the study

Patients listed for a deceased donor transplant will not be excluded.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | up to 24 weeks

SECONDARY OUTCOMES:
Diastolic Blood Pressure | up to 24 weeks
Treatment Costs | up to 24 weeks
Quality of Life | up to 24 weeks
Adverse Events/Symptoms | up to 24 weeks
Bone Health | up to 24 weeks
Anemia | up to 24 weeks
Nutrition and Growth | up to 24 weeks
Echocardiogram measured left ventricular mass | every 3 months
School Performance | every 3 months
Inflammatory Markers | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L Laskin, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (2):
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- The Hospital for Sick Children, Toronto, Canada